CLINICAL TRIAL: NCT06167824
Title: Assessment of Predictive Role of [11C] Choline PET/CT on Survival in Prostate Cancer Patients With Biochemical Failure Without Androgen Deprivation Therapy
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: PETCT-CHOL-SURVIVAL-TREATMENT
Record Dates: First submitted 2023-11-29; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among all the patients who underwent PET/CT with choline at our Institute between 2004 and 2007 to restage the prostatic disease following biochemical recovery of the disease, in this retrospective study the patients previously treated with radical prostatectomy, who present a progressive increase in the PSA value in the absence of hormone therapy and of which there is knowledge of the main clinical and follow-up data, with particular attention to survival data.

The PET/CT study with Choline, being part of the normal standard diagnostic work-up of patients, was performed following the normal clinical protocol. With the retrospective analysis of the data, the time elapsed following the prostatectomy operation and the follow-up time after the Choline PET/CT study will be evaluated and patients who died due to prostate cancer will therefore be considered. Prostate cancer-specific survival, calculated as the interval between radical prostatectomy and death due to prostate cancer, will be used as the end point. The differences between prostate cancer-specific survival of patients with a positive choline PET/CT study and patients with a negative choline PET/CT study will be evaluated (log-rank test). Choline PET/CT will be considered positive if pathological findings with significant tracer uptake are identified. In the subpopulation of patients with a positive Choline PET/CT study, survival data will also be evaluated in relation to the site of positivity of the PET/CT study, in particular at the level of local recurrence, in the lymph node or skeletal site.

ELIGIBILITY:
Inclusion Criteria:

* patients previously treated with radical prostatectomy, with progressive increase in PSA value in the absence of hormonal therapy.

Exclusion Criteria:

* < 18 years patients

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: patients previously treated with radical prostatectomy, with progressive increase in PSA value in the absence of hormonal therapy and for whom there is knowledge of the main clinical and follow up data with particular attention to survival data.
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2014-06-19 (Actual); Primary Completion 2014-07-15 (Actual); Study Completion 2014-07-15 (Actual)

PRIMARY OUTCOMES:
PET/CT with coline in patients previously treated with radical prostatectomy. | 1 year
  Retrospective observational study with 302 patients with prostate cancer were considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No